CLINICAL TRIAL: NCT04682223
Title: Center for the Study of Aphasia Recovery (C-STAR): Telerehabilitation for Aphasia (TERRA)
Brief Title: Telerehabilitation for Aphasia (TERRA)
Acronym: TERRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH); Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Julius Fridriksson, Primary Investigator, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00105675; P50DC014664 (NIH)
Record Dates: First submitted 2020-12-18; First posted 2020-12-23 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Aphasia; Stroke; Stroke Rehabilitation
Keywords: aphasia; stroke; telerehabilitation; speech-language therapy
MeSH Terms: conditions — Aphasia; Stroke; Communication Disorders

STUDY DESIGN:
Intervention Model Description: To conduct a randomized controlled phase II trial aimed at testing whether aphasia therapy delivered by a remote SLP through videoconferencing (aphasia remote therapy; ART) is non-inferior to in-clinic therapy (I-CT).
Who Masked: Outcomes Assessor
Masking Description: Raters will be blind to study timepoint, assignment of ART or I-CT, and treatment type (semantically- or phonologically-focused).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aphasia Remote Therapy (ART) (Experimental): All participants in this group will receive 3 weeks of daily semantically-focused treatment (semantic feature analysis, semantic barrier task and verb network strengthening therapy) and 3 weeks of daily phonologically-focused treatment (phonological components analysis, phonological production task, phonological judgment task). Participants will be randomized to order of treatment.
  All treatment will be done remotely with a speech-language pathologist through an online platform using therapy applications. Participants will be provided with teletherapy kits (including an Internet hotspot if needed) to complete the therapy tasks.
  Interventions: Behavioral: Semantically-focused therapy tasks; Behavioral: Phonologically-focused therapy tasks
- In-Clinic Therapy (I-CT) (Active Comparator): All participants in this group will receive 3 weeks of daily semantically-focused treatment (semantic feature analysis, semantic barrier task and verb network strengthening therapy) and 3 weeks of daily phonologically-focused treatment (phonological components analysis, phonological production task, phonological judgment task). Participants will be randomized to order of treatment.
  All treatment will be done in person with a speech-language pathologist at the UofSC Aphasia Lab.
  Interventions: Behavioral: Semantically-focused therapy tasks; Behavioral: Phonologically-focused therapy tasks

INTERVENTIONS:
Behavioral: Semantically-focused therapy tasks — 1) Semantic feature analysis (SFA; Boyle & Coelho, 1995; Boyle, 2004). For each pictured stimulus the participant is prompted to name the picture. Then, s/he is encouraged to produce semantically related words that represent features similar to the target word. 2) Semantic barrier task. This approach includes features of the Promoting Aphasics' Communication Effectiveness (PACE; Davis & Wilcox,1985). The goal of the task is for one participant (e.g., person with aphasia) to describe each card so that the other participant (e.g., clinician) can guess the picture on the card. 3) Verb network strengthening therapy (VNeST; Edmonds et al., 2009; 2014) targets lexical retrieval of verbs and their thematic nouns. The objective of VNeST is for the participant to generate verb-noun associates with the purpose of strengthening the connections between the verb and its thematic roles.
Behavioral: Phonologically-focused therapy tasks — 1) Phonological components analysis task (PCA; Leonard et al., 2008). The participant first attempts to name a given picture and then to identify the phonological features of the target words. 2) Phonological production task focuses on the identification of phonological features of targeted, imageable nouns and verbs. It requires the participant to sort picture stimuli based on the number of syllables and then to identify a hierarchy of phonological features. Once each targeted feature is identified for the pair of words, the participant is required to blend the syllables/sounds together. 3) Phonological judgment task relies on computerized presentation of verbs and nouns where participants are required to judge whether pairs of words include similar phonological features (e.g. # of syllables, initial phonemes, final phonemes, rhyming).

SUMMARY:
Speech-language therapy is generally found to be helpful in the rehabilitation of aphasia. However, not all patients with aphasia have access to adequate treatment to maximize their recovery. The goal of this project is to compare the efficacy of telerehabilitation or Aphasia Remote Therapy (ART) to the more traditional In-Clinic Therapy (I-CT).

DETAILED DESCRIPTION:
Stroke is the leading cause of adult disability in the United States. One of the most debilitating impairments resulting from stroke is aphasia, a language disorder caused by damage to the left hemisphere of the brain. While evidence shows that aphasia therapy improves speech production and communicative quality of life in persons with chronic (>6 months) stroke-induced aphasia, the amount of therapy provided to patients in the United States is typically far less than what is probably necessary to maximize recovery. There are a few important reasons underlying this discrepancy. For example, considerable emphasis is placed on acute and subacute stroke recovery with less therapy focus on the chronic period, when recovery is usually slower. Also, access to rehabilitation services can be limited by the availability of providers (e.g., in rural regions) or by difficulties with transportation logistics related to disabilities and the physical sequelae of stroke. One way to increase access to aphasia therapy is to rely on telerehabilitation (a.k.a., aphasia remote therapy; ART). So far, telerehabilitation in stroke has primarily focused on physical therapy, with only a handful of smaller studies involving aphasia therapy. The purpose of this study is to compare aphasia therapy administered via ART to aphasia therapy administered in person (In-Clinic Therapy; I-CT). We will conduct the first phase II, non-inferiority trial of telerehabilitation for aphasia therapy that is exclusively administered by a speech-language pathologist. Participants with chronic aphasia will be randomized to either a telerehabilitation or aphasia remote therapy (ART) group or an in-clinic therapy (I-CT) group relying on the same therapy approach currently used in our ongoing POLAR study. The outcome measure will focus on speech production and combines correct naming on the Philadelphia Naming Test and correct words produced per minute (CWPM) during discourse. The primary endpoint is change in the outcome measure at 6 months compared to baseline. The non-inferiority margin will be set so that if ART leads to less than 50% improvement than the improvement following I-CT, it will be considered inferior for therapy delivery. Neuroimaging will be used to evaluate how aphasia is shaped by the stroke lesion in combination with residual brain integrity.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have sustained a left hemisphere ischemic or hemorrhagic stroke at least 12 months prior to enrollment.
2. Participants must primarily speak English for at least the past 20 years.
3. Participants must be capable of giving informed consent or indicating another to provide informed consent.
4. Participants must be between 21-80 years of age.
5. Participants must be magnetic resonance imaging (MRI) compatible (e.g., no metal implants, not claustrophobic) on a 3-Tesla (3T) scanner.

Exclusion Criteria:

1. Participants must not have previous neurological disease affecting the brain (e.g. history of traumatic brain injury).
2. Participants must not have severely limited speech production (severe unintelligibility) and/or auditory comprehension that interferes with adequate participation in the therapy provided (i.e., WAB-R Spontaneous Speech rating scale score of 0-1 or WAB-R Comprehension score of 0-1).
3. Participants must not have a history of stroke to the right hemisphere of the brain.
4. Participants must not have a bilateral, cerebellar or brainstem stroke.
5. Participants must not have anything that makes them be 3T MRI incompatible
6. Insufficient intelligible speech to provide accurate responses with discourse/naming.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Speech Production Outcome Score (SPOTS) | Compare baseline score to 6 month follow-up (after treatment) score.
  A composite measure of naming (items correct on the Philadelphia Naming Test (PNT; Roach et al., 1996) and discourse words per minute (WPM)

SECONDARY OUTCOMES:
Improvement in overall aphasia severity | Compare baseline score to 6 month follow-up (after treatment) score.
  As measured by the Western Aphasia Battery-Revised (WAB-R; Kertesz, 2007)
Improvement in quality of life | Compare baseline score to 6 month follow-up (after treatment) score.
  As measured by the Stroke Aphasia Quality of Life Scale-39 (SAQOL-39; Hilari et al., 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Julius Fridriksson, Ph.D., Principal Investigator — University of South Carolina
Locations (1):
- University of South Carolina Aphasia Lab, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD will be shared via WebDCU™, a web based clinical trial management system developed by the Data Coordination Unit at the Medical University of South Carolina.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: IPD will be shared within 1 year of completion of the study.
Access Criteria: IPD available upon request.
URL: https://dcu.musc.edu/

REFERENCES:
- [Background] Bak TH, Hodges JR. Kissing and dancing-a test to distinguish the lexical and conceptual contributions to noun/verb and action/object dissociation. Preliminary results in patients with frontotemporal dementia. Journal of Neurolinguistics. 2003; 16(2): 169-181.
- [Background] Breitenstein C, Grewe T, Floel A, Ziegler W, Springer L, Martus P, Huber W, Willmes K, Ringelstein EB, Haeusler KG, Abel S, Glindemann R, Domahs F, Regenbrecht F, Schlenck KJ, Thomas M, Obrig H, de Langen E, Rocker R, Wigbers F, Ruhmkorf C, Hempen I, List J, Baumgaertner A; FCET2EC study group. Intensive speech and language therapy in patients with chronic aphasia after stroke: a randomised, open-label, blinded-endpoint, controlled trial in a health-care setting. Lancet. 2017 Apr 15;389(10078):1528-1538. doi: 10.1016/S0140-6736(17)30067-3. Epub 2017 Mar 1. PMID 28256356
- [Background] Brady MC, Kelly H, Godwin J, Enderby P, Campbell P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2016 Jun 1;2016(6):CD000425. doi: 10.1002/14651858.CD000425.pub4. PMID 27245310
- [Background] Brady MC, Kelly H, Godwin J, Enderby P. Speech and language therapy for aphasia following stroke. Cochrane Database Syst Rev. 2012 May 16;(5):CD000425. doi: 10.1002/14651858.CD000425.pub3. PMID 22592672
- [Background] Boyle M. Semantic feature analysis treatment for anomia in two fluent aphasia syndromes. Am J Speech Lang Pathol. 2004 Aug;13(3):236-49. doi: 10.1044/1058-0360(2004/025). PMID 15339233
- [Background] Boyle M, Coelho CA. Application of semantic feature analysis as a treatment for aphasic dysnomia. American Journal of Speech-Language Pathology. 1995; 4(4): 913-919.
- [Background] Cho-Reyes S, Thompson CK. Verb and sentence production and comprehension in aphasia: Northwestern Assessment of Verbs and Sentences (NAVS). Aphasiology. 2012;26(10):1250-1277. doi: 10.1080/02687038.2012.693584. PMID 26379358
- [Background] Conners C, Connelly V, Campbell S, MacLean M, Barnes J. Conners' Continuous Performance Test. Multi-Health Systems, Inc. 2000.
- [Background] Davis JD. The Boston Cooking School Magazine of Culinary Science and Domestic Economics. Boston, MA: Boston Cooking-School Magazine. 1901.
- [Background] Davis A, Wilcox J. Adult Aphasia Rehabilitation: Applied Pragmatics. San Diego, CA: Singular. 1985.
- [Background] Dell GS, Schwartz MF, Martin N, Saffran EM, Gagnon DA. Lexical access in aphasic and nonaphasic speakers. Psychol Rev. 1997 Oct;104(4):801-38. doi: 10.1037/0033-295x.104.4.801. PMID 9337631
- [Background] Edmonds LA, Mammino K, Ojeda J. Effect of Verb Network Strengthening Treatment (VNeST) in persons with aphasia: extension and replication of previous findings. Am J Speech Lang Pathol. 2014 May;23(2):S312-29. doi: 10.1044/2014_AJSLP-13-0098. PMID 24687125
- [Background] Edmonds LA, Nadeau SE, Kiran S. Effect of Verb Network Strengthening Treatment (VNeST) on Lexical Retrieval of Content Words in Sentences in Persons with Aphasia. Aphasiology. 2009 Mar 1;23(3):402-424. doi: 10.1080/02687030802291339. PMID 19763227
- [Background] Fotiadou D, Northcott S, Chatzidaki A, Hilari, K. Aphasia blog talk: How does stroke and aphasia affect a person's social relationships? Aphasiology. 2014; 28(11): 1281-1300.
- [Background] Grimes N. Walt Disney's Cinderella. New York, NY: Random House. 2005.
- [Background] Hilari K, Byng S, Lamping DL, Smith SC. Stroke and Aphasia Quality of Life Scale-39 (SAQOL-39): evaluation of acceptability, reliability, and validity. Stroke. 2003 Aug;34(8):1944-50. doi: 10.1161/01.STR.0000081987.46660.ED. Epub 2003 Jul 10. PMID 12855827
- [Background] Howard D, Patterson K, Franklin S, Orchard-Lisle V, Morton J. Treatment of word retrieval deficits in aphasia. A comparison of two therapy methods. Brain. 1985 Dec;108 ( Pt 4):817-29. PMID 4075074
- [Background] Kay J, Lesser R, Coltheart M. PALPA: Psycholinguistic assessments of language processing in aphasia. New York, NY: Psychology Press. 2009.
- [Background] Kertesz A. Western Aphasia Battery-Revised. San Antonio, TX: Pearson. 2007.
- [Background] Lau M. Who made that? New York Times Magazine, June 7, 2013.
- [Background] Laver KE, Adey-Wakeling Z, Crotty M, Lannin NA, George S, Sherrington C. Telerehabilitation services for stroke. Cochrane Database Syst Rev. 2020 Jan 31;1(1):CD010255. doi: 10.1002/14651858.CD010255.pub3. PMID 32002991
- [Background] Leonard C, Rochon E, Laird, L. Treating naming impairments in aphasia: Findings from a phonological components analysis treatment. Aphasiology. 2008; 22(9): 923-947.
- [Background] Menn L, Ramsberger G, Estabrooks NH. A linguistic communication measure for aphasic narratives. Aphasiology. 1994; 8(4): 343-59.
- [Background] Monsell S. On the relation between lexical input and output pathways for speech. In: Language Perception and Production: Relationships between Listening, Speaking, Reading and Writing. Cognitive science series. Academic Press. 1987: 273-311.
- [Background] Parmanto B, Lewis AN Jr, Graham KM, Bertolet MH. Development of the Telehealth Usability Questionnaire (TUQ). Int J Telerehabil. 2016 Jul 1;8(1):3-10. doi: 10.5195/ijt.2016.6196. eCollection 2016 Spring. PMID 27563386
- [Background] Roach A, Schwartz MF, Martin N, Grewal RS, Brecher A. The Philadelphia Naming Test (PNT): Scoring and rationale. Clinical Aphasiology. 1996; 24: 121-134.
- [Background] Simmons-Mackie N, Worral L, Murray L, Enderby, P. The top ten: Best practice recommendations for aphasia. Aphasiology. 2016; 31(2): 1-21.
- [Background] Strand EA, Duffy JR, Clark HM, Josephs K. The Apraxia of Speech Rating Scale: a tool for diagnosis and description of apraxia of speech. J Commun Disord. 2014 Sep-Oct;51:43-50. doi: 10.1016/j.jcomdis.2014.06.008. Epub 2014 Jul 14. PMID 25092638
- [Background] Utianski RL, Duffy JR, Clark HM, Strand EA, Botha H, Schwarz CG, Machulda MM, Senjem ML, Spychalla AJ, Jack CR Jr, Petersen RC, Lowe VJ, Whitwell JL, Josephs KA. Prosodic and phonetic subtypes of primary progressive apraxia of speech. Brain Lang. 2018 Sep;184:54-65. doi: 10.1016/j.bandl.2018.06.004. Epub 2018 Jul 4. PMID 29980072
- [Background] Venkatesh V, Davis FD. A model of the antecedents of perceived ease of use: Development and test. Decision Sciences. 1996; 27(3): 451-481.
- [Background] Wechsler D. Wechsler adult intelligence scale-Fourth Edition (WAIS-IV). San Antonio,TX: NCS Pearson. 2008.
- [Background] Winkler M, Bedford V, Northcott S, Hilari H. Aphasia blog talk: How does stroke and aphasia affect the carer and their relationship with the person with aphasia? Aphasiology. 2014; 28(11): 1301-1319.